CLINICAL TRIAL: NCT02634970
Title: CANadian Study in Patients With Wet AMD, Evaluating the Efficacy and Safety of Switching From Intravitreal Aflibercept to RanIbizumab
Acronym: CANARI
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002ACA09
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Wet Age-related Macular Degeneration (Wet AMD)
Keywords: wet AMD, ranibizumab, aflibercept, neovascularization
MeSH Terms: conditions — Neovascularization, Pathologic | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranibizumab at 0.5 mg (Experimental): Single arm, intravitreal injection
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 0.5 mg, intravitreal injection

SUMMARY:
There are limited prospective data regarding the potential benefit and risks associated with switching between anti-VEGF therapies in patients with nAMD who have initially achieved a favorable response to the first anti-VEGF therapy used but subsequently have evidence of increasing disease activity despite continuation of therapy. This study will fill this knowledge gap by prospectively evaluating the effectiveness and safety of switching from aflibercept to ranibizumab in nAMD patients that have non - sustained response to initial treatment with aflibercept.

ELIGIBILITY:
Inclusion Criteria:

* BCVA ≥23 ETDRS letters in study eye at both the Screening and Baseline visits.
* Evidence, at Screening, of active, angiographically confirmed Choroidal Neovascularization (CNV) secondary to AMD, directly or indirectly affecting the center of the fovea in study eye.
* No prior anti-VEGF treatment other than aflibercept.

Exclusion Criteria:

* History of cerebrovascular accident, transient ischemic attack or myocardial infarction within 3 months of the Screening visit.
* Any type of systemic disease or its treatment, including any medical condition (controlled or uncontrolled) that could be expected to progress, recur, or change to such an extent that it may bias the assessment of the clinical status of the patient to a significant degree or put the patient at special risk.

Exclusion criteria for ocular medical history and conditions for either eye:

* Any active periocular or ocular infection, or active intraocular inflammation at the time of Screening or Baseline (as per contraindications in the Lucentis® Product Monograph).
* Uncontrolled glaucoma (intraocular pressure [IOP] ≥30 mm Hg on medication or according to Investigator's judgment) at the time of Screening or Baseline
* Evidence of bilateral active CNV during the Screening Period or at Baseline requiring bilateral anti-VEGF injections.
* Prior intravitreal injection of ranibizumab or bevacizumab into the study eye and/or prior intravitreal injection of bevacizumab into the fellow eye.

Study eye exclusion criteria:

* At Baseline, intraocular surgery was performed within the previous 28 days or intraocular surgery is planned at any time during the 6 month study period
* Cataract (if causing significant visual impairment), aphakia, severe vitreous hemorrhage, rhegmatogenous retinal detachment, proliferative retinopathy or choroidal neovascularization of any other cause than wet AMD (e.g. ocular histoplasmosis, pathologic myopia (≥-8 dioptres)) at the time of Screening and Baseline.
* Irreversible structural damage involving the center of the fovea (e.g. advanced fibrosis or geographic atrophy) which in the opinion of the Investigator is sufficient to irreversibly impair visual acuity.
* Polypoidal choroidal vasculopathy (PCV), RPE tear, central serous retinopathy (CSR), or significant vitreomacular traction identified during Screening period or within 4 months of Baseline visit. Note that small vitreomacular adhesions that do not result in deformity of the retina are permitted.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Mean change in Central Subfield Retinal Thickness (CSRT) | at Day 90 (Month 3) and Day 180 (Month 6)
  Change (in absolute and percentage terms) in central subfield retinal thickness (CSRT) measured by spectral domain/ high definition optical coherence tomography (SD/HD-OCT).

SECONDARY OUTCOMES:
Mean change in Central Subfield Retinal Thickness (CSRT) | Monthly, from baseline to Month 6
  Change (in absolute and percentage terms) in central subfield retinal thickness (CSRT) measured by spectral domain/ high definition optical coherence tomography (SD/HD-OCT).
Mean change in Subfoveal Retinal Thickness (SRT) | Monthly, from baseline to Month 6
  Change (in absolute and percentage terms) in subfoveal retinal thickness (SRT) measured by spectral domain/ high definition optical coherence tomography (SD/HD-OCT).
Change in Central Subfield Retinal Volume (CSRV) | Monthly, from baseline to Month 6
  Change (in absolute and percentage terms) in subfoveal retinal thickness (SRT) measured by spectral domain/ high definition optical coherence tomography (SD/HD-OCT).
Mean change in Subretinal Fluid (SF) | Monthly, from baseline to Month 6
  Measured through Optical Coherence Tomography (OCT).
Mean change in Intra-Retinal Cystoid changes (IRCs) volume | Monthly, from baseline to Month 6
  Measured through Optical Coherence Tomography (OCT).
Mean change in Pigment Epithelial Detachments (PEDs) | Monthly, from baseline to Month 6
  Measured through Optical Coherence Tomography (OCT).
Mean change of Best-Corrected Visual Acuity (BCVA) | Monthly, from baseline to Month 6
  Best-corrected visual acuity (BCVA) will be assessed in a sitting position using subjective refraction and ETDRS-like visual acuity testing charts.
Rate of change in Subfoveal Retinal Thickness (SRT) | Monthly, from baseline to Month 6
  Rates will be assessed with the proportion of patients with changes.
Rate of change in Central Subfield Retinal Thickness (CSRT) | Monthly, from baseline to Month 6
  Rates will be assessed with the proportion of patients with changes.
Rate of change in Intra-Retinal Cystoid (IRCs) | Monthly, from baseline to Month 6
  Rates will be assessed with the proportion of patients with changes.
Rate of change in Pigment Epithelial Detachments (PEDs) | Monthly, from baseline to Month 6
  Rates will be assessed with the proportion of patients with changes.
Rate of Dry Retina | Monthly, from baseline to Month 6
  Rates will be assessed with the proportion of patients with changes.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Novartis Pharmaceuticals